CLINICAL TRIAL: NCT04268420
Title: Phase 1 Clinical Trial With Controlled Human Malaria Infection (CHMI) for Safety, Protective Efficacy, and Immunogenicity of Plasmodium Falciparum Malaria Protein (FMP013) Administered Intramuscularly With ALFQ Healthy Malaria-Naïve Adults
Brief Title: A Trial For The Study of Falciparum Malaria Protein 013 Administered Via Intramuscular Injection in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-19-04
Record Dates: First submitted 2020-02-04; First posted 2020-02-13 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Vaccine Reaction
Keywords: Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - "Low" Dose (Active Comparator): Part A vaccinees in the "low dose" arm will receive the lower dosing (20 μg FMP013 per 0.5 mL ALFQ) approximately 2 weeks prior to each vaccination. Vaccination to be delivered on 0,1,2 month.
  Interventions: Drug: FMP013; Drug: ALFQ
- Part A - "High" Dose (Active Comparator): Part A vaccinees in the "high dose" arm will receive the lower dosing (40 μg FMP013 per 1.0 mL ALFQ) approximately 2 weeks prior to each vaccination.
  Vaccination to be delivered on 0,1,2 month.
  Interventions: Drug: FMP013; Drug: ALFQ
- Part B - "Standard" Dose (Active Comparator): Part B vaccinees in the "high dose" arm will receive the lower dosing (40 μg FMP013 per 1.0 mL ALFQ) approximately 2 weeks prior to each vaccination.
  Vaccination to be delivered on 4,5,6 month.
  Interventions: Drug: FMP013; Drug: ALFQ
- Part B - "Delayed" Dose (Active Comparator): Part B vaccinees in the "high dose" arm will receive the lower dosing (40 μg FMP013 per 1.0 mL ALFQ) approximately 2 weeks prior to each vaccination.
  Vaccination to be delivered on 0,1,6 month.
  Interventions: Drug: FMP013; Drug: ALFQ
- Part B - "Delayed Fractional" Dose (Active Comparator): Part B vaccinees in the "high dose" arm will receive the lower dosing (40 μg FMP013 per 1.0 mL ALFQ) approximately 2 weeks prior to each vaccination.
  Vaccination to be delivered on 0,1,6 month.
  Interventions: Drug: FMP013; Drug: ALFQ
- Control (No Intervention): Up to 6 subjects will be enrolled (defined as receiving malaria challenge) later in the trial to serve as challenge controls. Additional subjects may be recruited as alternates to ensure that 6 control subjects undergo the challenge. Any alternates not challenged will be released from the study at day of challenge.

INTERVENTIONS:
Drug: FMP013 — Falciparum Malaria Protein-13
  Arms: Part A - "High" Dose; Part A - "Low" Dose; Part B - "Delayed Fractional" Dose; Part B - "Delayed" Dose; Part B - "Standard" Dose
Drug: ALFQ — ALF with QS-21, saponin molecule derived from the tree bark of Quillaja species
  Arms: Part A - "High" Dose; Part A - "Low" Dose; Part B - "Delayed Fractional" Dose; Part B - "Delayed" Dose; Part B - "Standard" Dose

SUMMARY:
A Phase 1, open label clinical study to evaluate the safety, immunogenicity, tolerability and efficacy of Plasmodium falciparum Malaria Protein 013 (FMP013) combined with (ALF with QS-21), saponin molecule derived from the bark of Quillaja species (ALFQ)) in healthy adult volunteers at different doses and dosing schedules.

DETAILED DESCRIPTION:
This is an open-label immunization with Controlled Human Malaria Infection (CHMI) study. Healthy, malaria-naïve adults, aged 18-55 years old will be recruited into one of 5 experimental cohorts in 2 parts.

In Part A, 2 experimental cohorts of 5 subjects each will receive a series of 3 vaccinations at 0, 1, and 2 months at 2 doses (the "low dose" arm and the "high dose" arm).

In Part B, 3 experimental cohorts of 10 subjects will receive a series of 3 vaccinations at 0, 1, 6 months (called the "delayed dose" arm), the "delayed fractional dose" arm is vaccinated at 0, 1, and 6 months with the 6 month dose being 1/5 the other doses, and the "standard" arm" at the 4th, 5th, and 6th month (after the first 2 vaccinations of the other 2 arms in Part B).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages 18-55 (inclusive);
2. Able and willing to provide written, informed consent;
3. Able and willing to comply with all research requirements, in the opinion of the Investigator;
4. Agreement to refrain from blood donation during the course of the study. Volunteers who have undergone CHMI can donate to other research once the study is complete but cannot donate to the American Red Cross for at least 3 years after the CHMI event;
5. Laboratory Criteria within 90 days before enrollment:

   * Hemoglobin ≥ 11.7 g/dL for women; ≥ 12.0 g/dL for men;
   * White Blood Cell count = 3,800-10,800 cells/mm3;
   * Platelets = 140,000-400,000/mm3;
   * Alanine aminotransferase (ALT; SGPT) 9-46 U/L male and 6-29 U/L female;
   * Serum creatinine ≤ 1.5 mg/dL;
   * Negative HIV testing (HIV Ab / antigen 4th generation screen with reflex confirmatory RNA testing);
   * Negative hepatitis B surface antigen (HBsAg) and hepatitis C antibody testing; Note: As above, Grade 1 lab abnormalities detected on screening may be repeated at PI discretion. Persistent Grade 1 abnormalities that are felt to represent the non-pathologic baseline for the subject will be discussed with the research monitor and documented before a subject is enrolled in the trial, and are allowable per discretion and agreement of the PI and Research Monitor
6. Birth control requirements:

   Female subjects must meet one of the following 2 criteria:
   * No reproductive potential due to post-menopausal status (12 months of natural [spontaneous] amenorrhea) or hysterectomy, bilateral oophorectomy or tubal ligation;
   * Women of childbearing potential should agree to practice highly effective contraception at least 30 days before enrollment and through 3 months post-CHMI or post-last vaccination (whichever is latest), using one of the following methods: condoms (male or female) with spermicide; diaphragm, or cervical cap with spermicide; intrauterine device; contraceptive pills, patch, injection, intravaginal ring or other FDA-approved contraceptive method; male partner has previously undergone a vasectomy; abstinence.

   Male subjects are encouraged but not required to practice highly effective contraception to avoid pregnancy in their partner from 30 days prior to enrollment through 60 days post-CHMI. This is due to the potential impact of malaria and antimalarial medications on spermatogenesis.
7. For all female subjects except those with a history of hysterectomy or bilateral oophorectomy, a negative β-HCG pregnancy test (urine) on day of enrollment, each day of vaccination, and the day of CHMI (tubal ligations have a not insignificant failure rate, 12 months of spontaneous amenorrhea does not completely preclude pregnancy and can be a result of polycystic ovarian syndrome);
8. Reachable (24/7) by mobile phone or other method of communication (email, landline, etc) during the period between CHMI and 28 days post-CHMI, per volunteer report;
9. No plans to travel outside the Washington DC metro area (DC, Maryland, and Virginia) between the day of challenge and 28 days post-challenge; For Travel outside the US occurring 28 days post-challenge to a malaria endemic area inclusion will be at the discretion of the PI.
10. If a subject is active duty military, he or she must obtain approval from his or her supervisor per WRAIR Policy 11-45;
11. Must have low (< 10%) cardiac risk factors according to clinical Gaziano (NHANES I) criteria assessed at screening, and a normal or normal variant ECG;
12. Completion of Study Comprehension Quiz (minimum passing score of 80% with 2 attempts permitted).
13. Subject must be willing to take anti-malarial treatment after CHMI;
14. Subject must provide 2 emergency contacts who will be made aware of the subject's participation in this trial and the vital importance of being reached during the challenge phase of the study. Both contacts must be verified by pone prior to subject enrollment.

Verification will be define as either speaking to the emergency contact over the phone, hearing their name included in the voicemail response, or confirming the emergency contact uses the number if a third party answers the phone.

Exclusion Criteria:

1. History of malaria infection (any species) or residence in a malaria-endemic area for more than 5 years (includes previous participation in CHMI studies).
2. Previous travel to malaria endemic regions within the past 6 months before study enrollment defined as first vaccination or day of challenge (for infectivity controls) or planned travel to malaria endemic regions during the vaccination, CHMI and 28-day CHMI follow-up period; For Travel outside the US occurring 28 days post-challenge to a malaria endemic area exclusion will be at the discretion of the PI.
3. Any history of receiving a malaria vaccine.
4. Received an investigational product in the 30 days before enrollment, or planned to receive during the study period.
5. Concurrent participation in another clinical research study.
6. Any use of medications that prevent or treat malaria during the 1 month prior to challenge or planned use during the study (outside of the drugs provided by the study team).
7. Any serious medical illness or condition involving the heart, liver, lungs, or kidneys.
8. Any significant risk for developing heart disease in the next 5 years, assessed according to clinical Gaziano (NHANES I) criteria assessed at screening, and an ECG.
9. Receipt of immunoglobulins or blood products within 3 months before enrollment.
10. Any history of anaphylaxis.
11. History of sickle cell trait or disease, or any condition that could affect susceptibility to malaria infection, per subject verbal report.
12. Pregnancy, lactation, or intention to become pregnant during the study, and 3 months after malaria challenge, if applicable.
13. Contraindications or allergies to the use of all 3 proposed anti-malarial medications; Malarone (atovaquone/proguanil), Coartem (artemether/lumefantrine) and chloroquine; contraindication to 1 or 2 is not exclusionary.
14. History of active/recent cancer still within treatment or active surveillance follow-up (except basal cell carcinoma of the skin and cervical carcinoma in situ). Treated/resolved cancers with no likelihood of recurrence may be deemed acceptable at Principal investigator discretion
15. History of autoimmune disease.
16. Significant (eg systemic anaphylaxis) hypersensitivity reactions to mosquito bites (local reactions at the site of mosquito bites are not an exclusion criterion) requiring hospitalization.
17. Suspected or known current alcohol or drug abuse as defined by an alcohol intake of greater than 3 drinks a day on average for a man, and greater than 2 drinks a day on average for a woman.
18. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to give informed consent, participate in the study, or impair interpretation of the study data, in the opinion of the Investigator.
19. Current anti-tuberculosis prophylaxis or treatment.
20. History of splenectomy.
21. History of confirmed or suspected immunodeficiency.
22. History of Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
23. History of Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years.
24. History of Diabetes mellitus (type I or II), with the exception of gestational diabetes.
25. History of Thyroid disease (except for well controlled hypothyroidism).
26. History of Idiopathic urticaria within the past year.
27. History of hypertension that is not well controlled by medication or that is persistently greater than 150/95 at screening...
28. History of bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
29. History of chronic or active neurologic disease to include seizure disorder and chronic migraine headaches. Exceptions are: i) childhood febrile seizures, or ii) seizures secondary to alcohol withdrawal more than 3 years ago.
30. Subjects receiving any of the following substances:

    * Systemic immunosuppressive medications or cytotoxic medications within 12 weeks before enrollment [with the exception of a short course of corticosteroids (≤ 14 days duration or a single injection) for a self-limited condition at least 2 weeks before enrollment; inhaled, intranasal or topical steroids are not considered exclusionary]
    * Treatment with known immunomodulators (other than nonsteroidal anti-inflammatory drugs [NSAIDs]) for any reason.
    * History of receipt of medication that prevent or treat malaria within 1 month of CHMI
    * Live attenuated vaccines within 30 days before initial study vaccine administration
    * Medically indicated subunit or killed vaccines, eg, influenza, pneumococcal, or allergy treatment with antigen injections, planned for administration 14 days before or after study vaccine administration
31. History of arthritis diagnosis other than osteoarthritis.
32. History of other diagnosed rheumatoid disorders.
33. Any history of psoriasis (itchy skin rash) or porphyria (rare disturbance of metabolism), since these conditions could get worse after treatment with chloroquine (a medication for treating malaria).
34. Subject must not have a fever in order to receive the study vaccine or participate in the malaria challenge.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety Dosage of Candidate Malaria Vaccine FMP013/ALFQ | 393 Days (+/-14)
  To assess the safety of candidate malaria vaccine FMP013/ALFQ. Safety dosage as indicated by incidence of solicited adverse events and serious adverse events through the end of the study.
Assess Reactogenicity of Candidate Malaria Vaccine FMP013/ALFQ | 393 Days (+/-14)
  To assess reactogenicity of candidate malaria vaccine. Occurrence of solicited local and systemic reactogenicity to FMP013/ALFQ

SECONDARY OUTCOMES:
Determine the Protective Efficacy of FMP013/ALFQ against a Plasmodium falciparum controlled human malaria infection. | 505 Days (+/-14)
  Proportion of vaccinated subjects without P.falciparum parasitemia (defined as one positive qRT-PCR test. Time to onset of P. falciparum parasitemia (defined as one positive qRT-PCR test) following CHMI.
Measure Immune Responses to CSP, induced by FMP013/ALFQ using various immunoassays. | 505 Days (+/-14)
  The Quantitative Anti-CSP IgG antibody titers, isotypes, and avidity measured by ELISA, ELISpot, and multiplex-based detection systems. Assess cellular immune responses to CSP by multicolor flow cytometry, ELISpot, and stimulation assays.
Measure Immune Responses to CSP, induced by FMP013/ALFQ using various immunoassays. | 505 Days (+/-14)
  The Qualitative Anti-CSP IgG antibody titers, isotypes, and avidity measured by ELISA, ELISpot, and multiplex-based detection systems. Assess cellular immune responses to CSP by multicolor flow cytometry, ELISpot, and stimulation assays.

OTHER OUTCOMES:
Compare the efficacy of standard, delayed dosing, and delayed fractional dosing | 505 Days (+/-14)
  Proportion of vaccinated subjects without P. falciparum parasitemia (defined as one positive qRT-PCR test and/or one positive TBS, whichever is first) following CHMI. Comparisons will be made across treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- WRAIR, Clinical Trials Center, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hutter JN, Robben PM, Lee C, Hamer M, Moon JE, Merino K, Zhu L, Galli H, Quinn X, Brown DR, Duncan E, Bolton J, Zou X, Angov E, Lanar DE, Rao M, Matyas GR, Beck Z, Bergmann-Leitner E, Soisson LA, Waters NC, Ngauy V, Regules J, Dutta S. First-in-human assessment of safety and immunogenicity of low and high doses of Plasmodium falciparum malaria protein 013 (FMP013) administered intramuscularly with ALFQ adjuvant in healthy malaria-naive adults. Vaccine. 2022 Sep 22;40(40):5781-5790. doi: 10.1016/j.vaccine.2022.08.048. Epub 2022 Aug 31. PMID 36055874

DOCUMENTS (3):
  • Informed Consent Form: Informed Consent Form Part B: C-D and C-F (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04268420/ICF_000.pdf
  • Informed Consent Form: Informed Consent Form Part B: Controls (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04268420/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form Part B: C-S (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04268420/ICF_002.pdf